CLINICAL TRIAL: NCT06757738
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1, Dose Escalation (With Optional Food Effect) Study of Orally Administered TRX-100 to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of TRX-100 in Healthy Volunteers
Brief Title: A Clinical Study Aiming to Assess Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of TRX-100 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TRX-100-0001; CT-2024-CTN-03164 (Other: therapeutic goods administration)
Record Dates: First submitted 2024-12-16; First posted 2025-01-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 4 cohorts (8 participant per cohort) to receive study drug
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single dose level 1 or placebo (Experimental): SAD dose level 1
  Interventions: Drug: TRX-100; Drug: Placebo
- Single dose level 2 or placebo (Experimental): SAD dose level 2
  Interventions: Drug: TRX-100; Drug: Placebo
- Single dose level 3 or placebo (Experimental): SAD dose level 3
  Interventions: Drug: TRX-100; Drug: Placebo
- Single dose level 4 or placebo (Experimental): SAD dose level 4
  Interventions: Drug: TRX-100; Drug: Placebo

INTERVENTIONS:
Drug: TRX-100 — CEN inhibitor, dosage form - capsules, dosing regimen - QD
Drug: Placebo — Placebo, dosage form - capsules, dosing regimen - QD

SUMMARY:
This is a clinical study aiming to assess pharmacokinetics, pharmacodynamics and preliminary efficacy of TRX-100 (and its major active metabolite TRX-101) in Healthy Volunteers

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled, dose escalation study to evaluate the safety, tolerability, PK, PD of orally administered TRX-100 (and its major active metabolite TRX-101) in Healthy Volunteers. The study will be conducted in 1 part only, as a single ascending dose (SAD) study at up to 4 dose levels. Evaluation of dose levels will be conducted in a sequential fashion with lower dose levels evaluated first in the sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 64 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg at screening.
4. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit and prior to dosing at the timepoints indicated in the SoA, including:

   1. Physical examination without any clinically significant findings in the opinion of the Investigator.
   2. Systolic blood pressure in the range of 90 mm Hg to 149 mm Hg; diastolic blood pressure in the range of 50 mm Hg to 90 mm Hg after 5 minutes in a supine or semi-supine position
   3. Heart rate (HR) in the range of 40 to 100 bpm
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.5°C (inclusive).
   5. No clinically significant findings in serum chemistry, hematology, coagulation and urinalysis tests as judged by the Investigator.
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine or semi-supine for at least 5 minutes) with a QTcF ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities.
   7. Hemoglobin A1C (HbA1c) levels within the local laboratory standard reference range.
5. Be willing to not smoke (including tobacco, nicotine replacement therapy, e-cigarettes) from 7 days prior to dose administration on Day 1 to Day 12 (inclusive) for all cohorts. For optional Cohort 4 only, participants must also be willing to not smoke (including tobacco, nicotine replacement therapy, e-cigarettes) from 7 days prior to dose administration on Day 28 to Day 39 (inclusive) .
6. Female volunteers must:

   1. Be of nonchildbearing potential i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause, and if under the age of 55 years a follicle-stimulating hormone (FSH) level >40 IU/L at the screening visit), or
   2. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from signing the consent form until at least 30 days after the last dose of the study drug.
7. Male volunteers, if not surgically sterilized, must agree to:

   1. Not donate sperm after signing consent, during the study, and at least 90 days after the EoS visit.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from signing the consent form until at least 90 days after the last dose of study drug.
8. Have suitable venous access for blood sampling.
9. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant.
2. Acute infections within 4 weeks prior to screening or current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the PI may affect absorption, distribution, metabolism or elimination of the study drug.
4. Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
5. Any screening laboratory result outside the normal laboratory reference range (as confirmed upon repeated testing) and deemed clinically significant by the PI.
6. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
7. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids by any route, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 5 half-lives of individual agent or within 28 days (whichever is longer) prior to Screening.
8. Use of or plans to use agents (e.g., grapefruit and grapefruit products) that have clinically significant interaction with CYP3A4 or the use of any medications that could have a significantly impact on organ function (e.g., barbiturates, omeprazole, cimetidine) during the study or within 5 half-lives of individual agent or within 7 days (whichever is longer) prior to dosing.
9. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or clinically significant arrythmia.
10. Participant is planning to have surgery between Screening and the EoS visit.
11. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies at the screening visit.
12. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
13. Estimated creatinine clearance < 60 mL/min using the Cockcroft-Gault formula.
14. Creatine kinase >2.0 x ULN at Day -1.
15. History of any drug or alcohol abuse in the past 2 years defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females. Where 1 unit = 360 mL of beer, 150 mL wine, or 30 mL of spirits.
16. History of alcohol consumption in the 48 hrs prior to dosing.
17. Positive drugs of abuse, or alcohol breath test results at the screening visit or at check-in (Day -1).
18. Use of any prescription medications within 14 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, including use of any over-the-counter medication (including herbal products, nutritional, diet aids, vitamin supplements, minerals) within 7 days or at least 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, with the exception of the occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days) or ibuprofen (doses of 400 mg up to every 6 hours or 1.2 g per day maximum for no more than 3 consecutive days), topical ointments, and vitamins or dietary supplements and medications used to manage AEs..
19. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
20. Known hypersensitivity to any of the study drug ingredients.
21. Use of any inactivated vaccinations within 14 days, or any live vaccinations within 30 days prior to the first study drug administration. Note: Participants vaccinated for COVID-19 or influenza within at least 2 weeks prior to enrollment or earlier will be considered eligible for enrollment as long as they do not present with post-vaccination clinical symptoms, have a negative rapid antigen test (in the case of COVID-19), and are deemed otherwise healthy.
22. For women of childbearing potential, a positive serum pregnancy test at the screening visit or a positive urine pregnancy test (with confirmatory serum pregnancy test) at check-in (Day -1).
23. Females who are breastfeeding or planning to breast feed at any time during the study.
24. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
25. Receiving an investigational drug in another clinical trial within 30 days or 5 half-lives of the investigational agent (whichever is longer) prior to the first study drug administration.
26. Any other condition or prior therapy that in the opinion of the Investigators would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
27. Any history of long COVID infection (defined by continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation).
28. Any history of severe influenza, defined as a confirmed diagnosis of influenza resulting in hospitalization, or symptoms severe enough to disrupt daily activities for more than 7 consecutive days.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Incidence, severity and relationship of AEs/serious AEs (SAEs) (including withdrawals due to AEs)
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Change from baseline in body weight in kg
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Change from baseline in systolic and diastolic blood pressure (mm Hg)
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Change from baseline in QRS duration (miliseconds)
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Change from baseline in heart rate (beats per minute)
To assess the safety and tolerability of a single oral administration of TRX-100 | up to Day 28
  Change from baseline in body temperature (Celsius)
To assess the safety and tolerability of a single oral administration of TRX-100 a | up to Day 28
  Change from baseline in QT interval (miliseconds)

SECONDARY OUTCOMES:
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Maximum observed concentration (Cmax)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Time to Cmax (Tmax)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUC0-last)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Area under the concentration-time curve from 0 to 24 hours (AUC0-24)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Area under the concentration-time curve from 0 to infinity (AUC0-inf)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Apparent terminal elimination half-life (t1/2)
To measure the pharmacokinetics of TRX-100 and its active metabolite TRX-101 in plasma | up to Day 28
  Terminal elimination rate constant (λz)

OTHER OUTCOMES:
Exploratory (optional): To evaluate TRX100/TRX101 target engagement. | up to Day 28
  • Inhibition of influenza virus replication in vitro measured as reduction on total plaques on Mason-darby canine kidney (MDCK) cell monolayers

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research, Sydney, Greater Sydney Area, Australia